CLINICAL TRIAL: NCT01322893
Title: Enumeration and Molecular Characterization of Circulating Tumour Cells in Women With Metastatic Breast Cancer
Acronym: CTC-MBC
Status: Completed | Type: Observational
Sponsor: Lund University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Version2. 2011-03-03
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Last update posted 2020-05-22 (Actual); Status verified 2019-05

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic breast cancer; Circulating tumour cells; CTC; Prognostic factors; Treatment response
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Blood sampling.: Blood samples will be taken before start of treatment, at month 1, month 3, month 4 and month 6.

SUMMARY:
Women with metastatic breast cancer, receiving first line treatment of any kind (chemotherapy, endocrine treatment or treatment with antibodies) will be included in this trial. In connection to treatment, blood samples for determination and enumeration of circulating tumour cells will be collected at different time points. Serum and plasma will be collected and stored for future analysis of RNA and DNA.

ELIGIBILITY:
Inclusion Criteria:

* Women with metastatic breast cancer
* ECOG performance status 0-2
* Age over18 years
* Signed informed concent
* Predicted life expectancy over 2 months
* Planned for first line systemic treatment for metastatic disease (chemotherapy, antibody treatment or endocrine treatment)
* Standard imaging evaluation within 4 weeks of inclusion
* Planned for standard imaging within 16 weeks after start of therapy

Exclusion Criteria:

* Prior medical therapy for metastatic disease (prior adjuvant chemotherapy, radiotherapy or endocrine therapy is permitted)
* Inability to understand information about the study
* Other malignant disease with the exception of curatively treated basal cell or squamous cell cancer of the skin and cancer in situ of the cervix

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with metastatic breast cancer
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2011-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
To determine whether numbers of circulating tumour cells in peripheral blood can give information of prognosis, and to evaluate if the numbers of circulating tumour cells can give information of the efficacy of given treatment | Blood samples will be taken before start of treatment, at month 1, month 3, month 4 and month 6.

CONTACTS AND LOCATIONS:
Locations (1):
- Lund University Hospital, Lund, Sweden

REFERENCES:
- [Derived] Gunnarsdottir FB, Bendahl PO, Johansson A, Benfeitas R, Ryden L, Bergenfelz C, Larsson AM. Serum immuno-oncology markers carry independent prognostic information in patients with newly diagnosed metastatic breast cancer, from a prospective observational study. Breast Cancer Res. 2023 Mar 21;25(1):29. doi: 10.1186/s13058-023-01631-6. PMID 36945037
- [Derived] Narbe U, Bendahl PO, Aaltonen K, Ferno M, Forsare C, Jorgensen CLT, Larsson AM, Ryden L. The Distribution of Circulating Tumor Cells Is Different in Metastatic Lobular Compared to Ductal Carcinoma of the Breast-Long-Term Prognostic Significance. Cells. 2020 Jul 17;9(7):1718. doi: 10.3390/cells9071718. PMID 32709042
- [Derived] Larsson AM, Jansson S, Bendahl PO, Levin Tykjaer Jorgensen C, Loman N, Graffman C, Lundgren L, Aaltonen K, Ryden L. Longitudinal enumeration and cluster evaluation of circulating tumor cells improve prognostication for patients with newly diagnosed metastatic breast cancer in a prospective observational trial. Breast Cancer Res. 2018 Jun 8;20(1):48. doi: 10.1186/s13058-018-0976-0. PMID 29884204
- [Derived] Jansson S, Bendahl PO, Larsson AM, Aaltonen KE, Ryden L. Prognostic impact of circulating tumor cell apoptosis and clusters in serial blood samples from patients with metastatic breast cancer in a prospective observational cohort. BMC Cancer. 2016 Jul 8;16:433. doi: 10.1186/s12885-016-2406-y. PMID 27390845
- [Derived] Frithiof H, Welinder C, Larsson AM, Ryden L, Aaltonen K. A novel method for downstream characterization of breast cancer circulating tumor cells following CellSearch isolation. J Transl Med. 2015 Apr 21;13:126. doi: 10.1186/s12967-015-0493-1. PMID 25896421
- See also: A novel method for downstream characterization of breast cancer circulating tumor cells following CellSearch isolation. - PubMed - NCBI — https://www.ncbi.nlm.nih.gov/pubmed/25896421
- See also: Prognostic impact of circulating tumor cell apoptosis and clusters in serial blood samples from patients with metastatic breast cancer in a prospec... - PubMed - NCBI — https://www.ncbi.nlm.nih.gov/pubmed/27390845
- See also: A FISH-based method for assessment of HER-2 amplification status in breast cancer circulating tumor cells following CellSearch isolation. - PubMed - NCBI — https://www.ncbi.nlm.nih.gov/pubmed/27895501
- See also: Evolution of Estrogen Receptor Status from Primary Tumors to Metastasis and Serially Collected Circulating Tumor Cells. — https://www.ncbi.nlm.nih.gov/pubmed/32326116
- See also: Serial evaluation of serum thymidine kinase activity is prognostic in women with newly diagnosed metastatic breast cancer. — https://www.ncbi.nlm.nih.gov//pubmed/32161278
- See also: Longitudinal CTC and CTC-cluster evaluation improves prognostication and monitoring in metastatic breast cancer patients during 1st line systemic treatment. — https://www.ncbi.nlm.nih.gov/pubmed/29884204
- See also: Prognostic impact of circulating tumor cell apoptosis and clusters in serial blood samples from patients with metastatic breast cancer in a prospective observational cohort. — https://www.ncbi.nlm.nih.gov/pubmed27390845
- See also: Molecular characterization of circulating tumor cells from patients with metastatic breast cancer reflects evolutionary changes in gene expression under the pressure of systemic therapy. — https://www.ncbi.nlm.nih.gov/pubmed/28489591
- See also: A FISH-based method for assessment of HER-2 amplification status in breast cancer circulating tumor cells following CellSearch isolation. — https://www.ncbi.nlm.nih.gov/pubmed/27895501
- See also: A novel method for downstream characterization of breast cancer circulating tumor cells following CellSearch isolation. — https://www.ncbi.nlm.nih.gov/pubmed/25896421